CLINICAL TRIAL: NCT06328361
Title: Nordic ORgan Preservation Pilot Approach - A Nonrandomised Single-Arm Trial for Non-Operative Management of Rectal Cancer (NORPPA-1)
Brief Title: Nordic ORgan Preservation Pilot Approach Nonrandomised Single-Arm Trial for Non-Operative Management of Rectal Cancer
Acronym: NORPPA-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other); Oulu University Hospital (Other); Jyväskylä Central Hospital (Other); Seinajoki Central Hospital (Other); Satakunta Central Hospital (Other); North Karelia Central Hospital (Other); Tartu University Hospital (Other); East Tallinn Central Hospital (Other); West Tallinn Central Hospital (Unknown); North Estonia Medical Centre (Other); Vaasa Central Hospital, Vaasa, Finland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R24008
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Organ Preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nonoperative management (Experimental): The patients presenting with complete clinical response undergo nonoperative management (i.e. watch & wait) as surveillance for local regrowth or distant spread.
  Interventions: Procedure: Nonoperative surveillance

INTERVENTIONS:
Procedure: Nonoperative surveillance — Clinical and imaging surveillance with digital rectal examination and/or endoscopy, rectal MRI and body CT
  Other Names: Watch and Wait; Organ preservation

SUMMARY:
The goal of this one-arm clinical trial is to implement and study the oncological outcomes of nonoperative management of rectal cancer having complete clinical response to neoadjuvant therapy. The main questions to answer are

* if the oncological results of nonoperative management after Nordic practice in chemoradiotherapy indications differ from experiences elsewhere
* what is the organ preservation rate
* what is the local regrowth rate

DETAILED DESCRIPTION:
Background: Non-operative management (NOM) for rectal cancer is an accepted treatment option that has not been commonly utilized in Finland but has been widely adopted in major cancer centers worldwide. NOM can be considered if the rectal tumor disappears with neoadjuvant treatment, resulting in a complete clinical response.

Objective: The aim of the study is to establish a unified NOM protocol for national use and determine whether the outcomes of Finnish and Estonian treatment practices align with international experiences.

Design: The study is a prospective, non-randomized, single-arm, international multicenter trial examining the oncological and quality-of-life consequences of NOM.

Primary Endpoint: The primary endpoint is disease-free survival 2 years after the initiation of NOM.

Secondary Endpoints: These include overall survival, disease-specific survival, survival free from total mesorectal excision (TME) surgery, survival free from circulating tumor DNA (ctDNA) detection after complete clinical response, recurrence-free survival, incidence of local recurrence and metastases, salvage TME success rate, quality of life at 1 year post-NOM, and treatment-related morbidity up to 5 years.

Inclusion Criteria: Patients must have histopathologically confirmed primary rectal adenocarcinoma before neoadjuvant treatment, achieve clinical complete response (cCR) after neoadjuvant therapy, and express willingness to undergo rectum-preserving treatment after considering the risk of recurrence.

Exclusion Criteria: Patients with evidence of metastasis at diagnosis, aged under 18, those not receiving neoadjuvant treatment, or those unable to provide informed consent are excluded.

Diagnosis and Treatment: Pretreatment of patients follows standard practice. Upon meeting inclusion criteria with confirmed cCR, patients undergo protocolized monitoring with clinical examination, laboratory tests, and imaging.

Randomization: No randomization is performed.

Follow-up: Patients are monitored every 3 months for the first 2 years, then every 6 months for 3 years. Monitoring replaces surgical intervention unless cancer recurs. Follow-up is part of standard care, with costs covered by the healthcare system.

Safety: Incidence of local recurrence and success of resection post-recurrence are monitored closely. If over 30% local recurrence occurs post-cCR, it may necessitate study termination at the center.

Data Collection: Clinical data are entered into electronic case report forms (eCRFs) based on primary healthcare documentation and stored pseudonymized on the primary research center's server. Molecular and pseudonymized clinical data are collected securely for analysis.

Sample Size Calculation and Statistical Analysis: A sample of 200 patients is estimated to provide sufficient data for the primary and key secondary endpoints and to meet other study objectives accurately.

Data Handling: Data handling adheres to privacy legislation, with information stored pseudonymously.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological verification of primary rectal adenocarcinoma
* Complete clinical response at response assessment after neoadjuvant therapy
* Informed consent to organ preservation study

Exclusion Criteria:

* Evidence of metastatic disease (fulfilling M-class criteria of TNM)
* No neoadjuvant therapy
* Inability to understand the information related to harms and benefits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  Survival from complete clinical response to locoregional failure or distant metastases

SECONDARY OUTCOMES:
Overall survival | 5 years
  Survival from complete clinical response to death or censoring of observation
TME-free survival | 5 years
  Survival from complete clinical response to total mesorectal excision surgery
ctDNA-free survival | 5 years
  Survival from complete clinical response to positive ctDNA result
Post local regrowth disease-free survival | 5 years
  Survival from operated local regrowth to recurrence
Post local regrowth overall survival | 5 years
  Survival from operated local regrowth to death or censoring of observation
Local regrowth-free survival | 5 years
  Survival from complete clinical response to local regrowth
Local recurrence-free survival | 5 years
  Survival from complete clinical response to local recurrence after local regrowth
Distant metastases-free survival | 5 years
  Survival from complete clinical response to distant metastases
Disease-free survival | 5 years
  Survival from complete clinical response to locoregional failure or distant metastases
Salvage rate after local regrowth | 5 years
  Rate of successful TME surgery, local excision or metastasectomy after local regrowth
Quality of life score | 5 years
  Baseline and change in quality of life after complete clinical response
Complication rates | 5 years
  Clavien-Dindo complications after NOM and after local regrowth and after recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Toni T Seppälä, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (13):
- Estonia (4):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Finland (9):
  - Helsinki University Central Hospital, Helsinki
  - Jyväskylä Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Seinajoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: No
The European Data Protection Regulation (GDPR) does not allow sharing other than anonymised patient level data.